CLINICAL TRIAL: NCT05412680
Title: Transoral Endoscopic Thyroidectomy by Vestibular Approach (TOETVA) Compared to Conventional Thyroidectomy by Cervical Approach: a Randomized Clinical Trial
Brief Title: Transoral Endoscopic Thyroidectomy by Vestibular Approach (TOETVA)
Acronym: TOETVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fábio de Aquino Capelli (Other)
Responsible Party: Sponsor-Investigator, Fábio de Aquino Capelli, Principal Investigator, Instituto do Cancer do Estado de São Paulo
Organization: Instituto do Cancer do Estado de São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOETVA
Record Dates: First submitted 2022-05-18; First posted 2022-06-09 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-03

CONDITIONS: Thyroid Diseases; Thyroid Cancer
MeSH Terms: conditions — Thyroid Diseases; Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TOETVA (Active Comparator): Patients submitted to transoral endoscopic thyroidectomy by vestibular approach
  Interventions: Procedure: TOETVA
- CONVENTIONAL THYROIDECTOMY (Active Comparator): Patients submitted to conventional open thyroidectomy by cervical approach
  Interventions: Procedure: conventional thyroidectomy

INTERVENTIONS:
Procedure: TOETVA — TRANSORAL ENDOSCOPIC THYROIDECTOMY BY VESTIBULAR APPROACH
  Arms: TOETVA
Procedure: conventional thyroidectomy — conventional open thyroidectomy by cervical approach
  Arms: CONVENTIONAL THYROIDECTOMY

SUMMARY:
Prospective study carried out with ICESP (instituto do Câncer do Estado de São Paulo) patients with thyroid disease with surgical indication

DETAILED DESCRIPTION:
Prospective study carried out with ICESP patients with thyroid disease with surgical indication, according to the aforementioned inclusion criteria, totaling 60 cases, which will be randomized into two groups:

* Conventional Thyroidectomy (30 patients)
* Transoral Endoscopic Thyroidectomy By Vestibular Approach (30 patients)

ELIGIBILITY:
Inclusion Criteria:

* history of hypertrophic scarring and/or motivation to avoid cervical scarring,
* maximum diameter of the thyroid < 10 cm and of the dominant nodule < 6 cm,
* estimated thyroid volume < 45 ml
* benign lesion (multinodular goiter, cyst),
* indeterminate nodule (Bethesda III or IV),
* suspicious nodule for well-differentiated thyroid carcinoma (Bethesda V and VI) < 2 cm

Exclusion Criteria:

* history of previous surgery or irradiation in the head and neck region and superior mediastinum
* evidence of clinical hyperthyroidism
* preoperative recurrent nerve palsy
* lymph node metastasis
* extra-thyroid extension
* plunging goiter
* oral abscess

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To compare TOETVA technique with conventional thyroidectomy in terms of operative time | 1 year
  Operative time will be measured by minutes
To compare TOETVA technique with conventional thyroidectomy in terms of post operative surgical complications, such as laryngeal nerve dysfunction | 1 year
  This outcome will be accessed by performing laryngoscopy before and after the surgery
To compare TOETVA technique with conventional thyroidectomy in terms of post operative surgical complications, such as hypoparathyroidism | 1 year
  This outcome will be accessed by accessing de blood calcium and parathormone levels after the surgery
To compare TOETVA technique with conventional thyroidectomy in terms of post operative surgical complications, such as hematoma formation | 1 year
  This outcome will be accessed by qualitative analysis
To compare TOETVA technique with conventional thyroidectomy in terms of post operative surgical complications, such as seroma formation | 1 year
  This outcome will be accessed by qualitative analysis
To compare TOETVA technique with conventional thyroidectomy in terms of post operative surgical complications, such as skin injury | 1 year
  This outcome will be accessed by qualitative analysis
To compare TOETVA technique with conventional thyroidectomy in terms of post operative pain | 1 year
  This outcome will be accessed by visual pain scale from grade 1 (better) to 10 (worse)
To compare TOETVA technique with conventional thyroidectomy in terms of time of hospitalization | 1 year
  This outcome will be accessed by number of days spent in the hospital

SECONDARY OUTCOMES:
Comparison on quality of life - questionnaire 1. | 1 year
  Quality of life evaluated by specific questionnaires, such as University of Washington version 4 - 0 (worse) 1200 (better)
Comparison on quality of life - questionnaire 2. | 1 year
  Quality of life evaluated by specific questionnaires, such as Dermatology life quality index - 0 (better) 30 (worse)
Comparison on quality of life - questionnaire 3. | 1 year
  Quality of life evaluated by specific questionnaires, such as Euroqol - 5D - 5 (better) 15 (worse)

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Capelli, phd, Principal Investigator — Instituto do Cancer do Estado de São Paulo
Locations (1):
- ICESP, São Paulo, São Paulo, Brazil